CLINICAL TRIAL: NCT05419037
Title: Natural History of Pregnancy and Pregnancy Outcomes in Metreleptin-Treated vs Untreated Subjects With Lipodystrophy
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000757; 000757-DK
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11-20

CONDITIONS: Lipodystrophy
Keywords: Metreleptin; Pregnancy; Off-Spring; Natural History
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- off-spring of above: Off-spring of the women who took metreleptin during her pregnancy.
- Women with past pregnancy on metreleptin: Women who took metreleptin during pregnancy.

SUMMARY:
Background:

Lipodystrophy is a health problem in which the body does not have enough fat tissue. People with lipodystrophy may not make enough of the hormone leptin. Leptin regulates hunger. Low leptin levels trigger hunger. People with lipodystrophy can have many health problems. They may take a drug (metreleptin) that mimics leptin. Little is known about how taking metreleptin may affect a pregnancy. Metreleptin may be helpful or harmful to pregnant women. It may also affect the health of the child who is born.

Objective:

This natural history study will collect data about the effects of taking metreleptin while pregnant.

Eligibility:

Women aged 18 years or older with lipodystrophy who have been pregnant. Women who did and who did not take metreleptin during their pregnancies are needed. Children of women with lipodystrophy who took this drug during pregnancy are also needed.

Design:

Participants will have 1 study visit. This visit may be by phone, by telehealth, or in-person.

Participants will answer questions about their pregnancies.

They will discuss any health problems they had.

They will be asked about any medicines they took before and during their pregnancies.

They will be asked about the health of their children.

Participants medical records will be reviewed.

Participants may need to provide a blood sample. They may also be asked to provide a sample of breastmilk.

Participants children may also be asked to provide a blood sample....

DETAILED DESCRIPTION:
Study Description:

Single-site cross-sectional study of women with lipodystrophy who had pregnancies during which they were or were not exposed to metreleptin, and the offspring of women whose offspring were exposed to metreleptin during pregnancy. The study involves secondary use of data and samples from other studies in which these subjects participated, review of outside medical records, and collection of a single blood specimen if a biobanked specimen is not available.

The hypotheses are:

1. Pregnancy complications will be less prevalent and severe in women with lipodystrophy who took metreleptin during pregnancy compared to those who did not, due the beneficial effects of metreleptin on metabolic complications of lipodystrophy.
2. Anti-leptin antibodies may be detected in some offspring born to women with lipodystrophy treated with metreleptin during pregnancy, but these antibodies will not be associated with adverse health outcomes.

Objectives:

Primary: Determine pregnancy outcomes, including type and frequency of pregnancy complications in women treated with metreleptin during pregnancy vs. untreated pregnancies.

Secondary: Determine if anti-leptin antibodies are detectable in offspring of women treated with metreleptin during pregnancy.

Endpoints:

Primary Endpoint: We will quantify a set of pregnancy and offspring outcomes and complications.

Secondary Endpoints: Frequency and type of anti-leptin antibodies.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Women with lipodystrophy who had pregnancies with or without use of metreleptin:

  * Female, aged >= 18 years
  * Clinical diagnosis of non-HIV associated generalized or partial lipodystrophy
  * History of one or more pregnancies
* Offspring of women with lipodystrophy who had pregnancies while taking metreleptin:

  * Males or females aged >=1 month
  * Mothers took metreleptin during their pregnancy
  * Availability of a biobanked blood specimen or willingness to provide a blood specimen

Note that subjects treated with metreleptin during pregnancy may participate in this study regardless of the participation of their offspring.

EXCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must not meet any of the following criteria:

* Inability of subject or guardian to understand or the unwillingness to sign a written informed consent document (except as noted below with *)
* Pregnancy.

  * Subjects who otherwise meet inclusion/exclusion criteria but who are not reachable to obtain informed consent may be included under a waiver of consent.

Ages: 6 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who were pregnant while taking metreleptin and their off-spring will be evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-07 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
type and frequency of pregnancy complications | at end of study
  We will quantify a set of pregnancy and offspring outcomes and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Result of the study will be disseminated to participants upon publication.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000757-DK.html